CLINICAL TRIAL: NCT04078750
Title: Pre-Transplant Multidisciplinary Assessment on Medication Adherence and Transplant Outcomes
Brief Title: PLATO - Medication Adherence in Transplant Recipients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, John Gill, Professor of Medicine, Division of Nephrology, Principal Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H19-02030
Record Dates: First submitted 2019-08-21; First posted 2019-09-06 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Kidney Disease, Chronic; Medication Adherence; Renal Disease; Kidney Rejection Transplant
MeSH Terms: conditions — Renal Insufficiency, Chronic; Medication Adherence; Kidney Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase I. Control group (Sham Comparator): 1. The standard of care will be provided to the control group pre- and post-transplant. This does not involve any direct pre-transplant assessment of medication adherence or risk factors for non-adherence.
  2. Tacrolimus capsules will be dispensed in Medication Event Monitoring System (MEMS) caps for 3 months post-transplant for the purpose of measuring adherence after transplantation.
  3. Patients will be asked to complete Basel Assessment of Adherence to Immunosuppressive Medication instrument (BAASIS) questionnaire and Long-term Medication Behaviour Self-efficacy Scale at 3 months after transplantation.
  Interventions: Behavioral: Tailored medication adherence plan
- Phase II. Intervention group (Experimental): Patients will be given lactose containing white- and yellow-colored gelatin capsules stored in (MEMS®) bottles for a 1-month adherence trial. Yellow-colored gelatin capsules represent tacrolimus 0.5mg capsules while white-colored gelatin capsules represent tacrolimus 1mg capsules. MEMS® is designed to record the date/time of opening and closure of the drug vial. Patients will be asked to take a certain dose and expected to remove the correct number of white and yellow capsules from respective vial at the correct time each day. Phone calls will be made to patients to change the 'dose' at various times throughout the month to mimic the frequent need to make tacrolimus dosing changes early post-transplant.Pill count and MEMS record will be reviewed at the end of the 1-month trial period to assess adherence. Patients will also undergo health literacy, cognition testing, self-efficacy tests, with a customized post-transplant plan.
  Interventions: Behavioral: Tailored medication adherence plan

INTERVENTIONS:
Behavioral: Tailored medication adherence plan — Comparison of mean daily medication adherence between intervention and control groups over 3 months, as measured by MEMS caps.

SUMMARY:
Non-adherence with immunosuppressant drugs is a major reason for premature kidney transplant failure. Currently, patient education and compliance aids (e.g bubble packing) are commonly used to assist patients. This is a study involving patients expected to undergo a kidney transplant within 6 months. One group will undergo a one-month formal assessment of adherence before transplantation using mock immunosuppressant medication. Standardized surveys will also be administered to assess risk factors for non-adherence. A plan will be developed for use after the transplant. The other group will undergo usual care. Kidney function and rejection rates will be compared between two groups.

DETAILED DESCRIPTION:
Phase I - Control group.

1. The standard of care will be provided to the control group pre- and post-transplant. This does not involve any direct pre-transplant assessment of medication adherence or risk factors for non-adherence.
2. Tacrolimus capsules (standard of care immunosupression medication) will be dispensed in Medication Event Monitoring System (MEMS) caps for 3 months post-transplant for the purpose of measuring adherence after transplantation.
3. Patients will be asked to complete Basel Assessment of Adherence to Immunosuppressive Medication instrument (BAASIS) self-report questionnaire and Long-term Medication Behaviour Self-efficacy self-report Scale at 3 months after transplantation.

Phase II - Interventional Group.

I. Pre-transplant phase:

1. Measurement of Adherence to Medications Patients will be given lactose containing white- and yellow-colored gelatin capsules stored in (MEMS®) bottles for a 1-month adherence trial. Yellow-colored gelatin capsules represent tacrolimus 0.5mg capsules while white-colored gelatin capsules represent tacrolimus 1mg capsules. MEMS® is designed to record the date/time of opening and closure of the drug vial. Patients will be asked to take a certain dose and expected to remove the correct number of white and yellow capsules from respective vial at the correct time each day. Phone calls will be made to patients to change the 'dose' at various times throughout the month to mimic the frequent need to make tacrolimus dosing changes early post-transplant. For patients who are lactose intolerance, they will be instructed to remove the correct number of capsules from the vials but there is no need to take the capsules. Pill count and MEMS record will be reviewed at the end of the 1-month trial period to assess adherence.
2. Health literacy: Assessments to completed by the participant:

   1. Short Literacy Survey (SLS), a self-report 3 question survey, has been validated in kidney transplant recipients and shown to correlate well with the Rapid Estimate of Adult Literacy in Medicine (REALM) and the shortened Test of Functional Health Literacy in Adults (S-TOFHLA). The three questions are: 1) "How often do you have someone help you read hospital materials?"; 2) "How confident are you filling out medical forms by yourself?"; and 3) "How often do you have problems learning about your medical condition because of difficulty understanding written information?"
   2. Newest Vital Signs - transplant version (NVS-T) The original NVS consists of a prescription label with 6 questions that measures health literacy and numeracy skills but is not specific to any particular area of medicine. The modified transplant version consists of 2 prescription labels and has been validated. The first label is for an antibiotic, amoxicillin, and the second label is for a cream, fluocinolone acetonide. There are 3 questions for each label, and the number of correct answers correlates with a health literacy category.
3. Cognition will be assessed using the Montreal Cognitive Assessment (MoCA), a 30-question screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
4. Self-efficacy will be assessed using the Long-term Medication Behaviour Self-efficacy Scale, a 27-item questionnaire about skills related to medication use. It assesses the following themes regarding patient's self-efficacy: personal attributions (7 items), environmental factors (13 items), task-related and behavioral factors (7 items).
5. Customized post-transplant care plan prior to transplantation The post-transplant team will devise a tailored care plan based on assessment findings and discussed with the patient and/or caregivers prior to transplant. The post-transplant care plans will be common to both transplant programs.

II. Post-transplant phase:

1. The post-transplant team will implement the tailored care plan as discussed with patient and/or caregiver(s).
2. Tacrolimus capsules will be dispensed in MEMS caps for 3 months post-transplant for the purpose of measuring adherence after transplantation.
3. Patients will be asked to complete BAASIS questionnaire and Long-term Medication Behaviour Self-efficacy Scale at 3 months.

Current standard of care does not include any element of pharmacy evaluation of a person's ability to follow medication regimens.

At the conclusion of the use of MEMS caps subjects in either group will return the MEMS caps to the pharmacists at a regularly scheduled follow-up appointment.This will not require an additional trip to the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant candidates anticipated to undergo transplantation from a deceased or living donor within 6 months of enrolment

Exclusion Criteria:

* There are no exclusion criteria. All eligible patients will be approached by a research assistant. Patients with limited English language fluency will be asked to participate with the assistance of a translator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of mean daily medication adherence between intervention and control groups over 3 months, as measured by MEMS caps. | 3 month duration
  Adherence is defined as patient opening the MEMS caps within 1 hour of dosing times (ie no missed doses AND ≤ 1-hour variations to scheduled dosing times). Assumption will be made that patient has taken the correct tacrolimus dose if he or she opens MEMS caps within predefined dosing times. Using the MEMS recorded electronic dosing history, a daily binary adherence rate will be calculated per patient (ie day with correct dosing and/or timing). It is recognized that adherence rate may wane over time post-transplant. A 3-month duration is chosen for the primary outcome for logistical reasons since out-of-town patients are usually transferred back to a peripheral transplant center closer to home at this time. A pilot will be conducted for 40 local transplant recipients (20 each in control and interventional groups) to extend the use of MEMS for 6 months to capture any differences in adherence rates beyond three months.

SECONDARY OUTCOMES:
Self-reported adherence rates as measured by BAASIS | 3-12 months
  Patients will be asked by research assistant to complete BAASIS questionnaire at 3 months after transplant (may be a phone call if patients are transferred to peripheral centers before 3 months).
The coefficient of variation (CV) of tacrolimus trough levels | 3-12 months
  The coefficient of variation (CV) of tacrolimus trough levels at 3 months and at 12 months will be assessed. We will compare the proportion of patients with CV ≥ 30% at 3 months and at 12 months. The 12-month measurement will be assessed in all patients including patients who receive care in peripheral transplant centers as this information is readily accessible in our electronic records. These measures will also help to address the long-term durability of any change in adherence related to the interventions.
Proportion of patients within target tacrolimus trough levels | 3-12 months
  Proportion of patients within target tacrolimus trough levels at 3 months and at 12 months.
Comparison of post-transplant test results between intervention and control group | 3 months
  Comparison of post-transplant test results between intervention and control group using a Long-term Medication Behaviour Self-efficacy Scale. The scale has 5 possible answers that reflect the extent that the participant is able to take their medications correctly in the described situations.
  1. unlikely
  2. maybe, maybe not
  3. probably yes
  4. most probably
  5. certainly
Medication Behaviour for intervention group only | 3 months
  Comparison of post-transplant test results between intervention and control group using a Long-term Medication Behaviour Self-efficacy Scale. The scale has 5 possible answers that reflect the extent that the participant is able to take their medications correctly in the described situations.
  1. unlikely
  2. maybe, maybe not
  3. probably yes
  4. most probably
  5. certainly
Staff resource utilization | Through study completion, an average of 1 year
  Time spent with patient education + re-education + discharge planning + resolving medication errors + arranging for medication management. The post-transplant team will receive an inservice to ensure accurate and complete documentation of their time spent on the above activities.
Medication nonadherence-related hospital readmissions | 12 months
  Medication nonadherence-related hospital readmissions will be assessed for 12 months after transplantation by review of all hospitalization records.
Biopsy proven acute rejection (BPAR) rate | 12 months
  Biopsy proven acute rejection (BPAR) rate at 12 months
Kidney allograft function | 12 months
  Kidney allograft function (SCr, UACR) at 12 months
Kidney allograft survival | 12 months
  Kidney allograft survival at 12 months
Patient survival | 12 months
  Patient survival at 12 months
Health Literacy for intervention group only | 3 months
  This group will also undergo health literacy surveys which associates answers with values of 1-5: A lower score indicates lower health literacy.
Montreal Cognitive Assessment for intervention group only | 3 months
  Cognition will be assessed using the Montreal Cognitive Assessment (MoCA), a 30-question screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Leung, Pharm D, Principal Investigator — St. Paul's Hospital
Locations (2):
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No